CLINICAL TRIAL: NCT00337272
Title: Phase IV: Treatment of Chronic Insomnia in Patients With Breast Cancer Following Completion of Chemotherapy
Brief Title: Treating Chronic Insomnia in Breast Cancer Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACORN AEJSINS0601
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Insomnia
Keywords: chronic insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo) (Placebo Comparator): Patients will take placebo 30 minutes before bedtime days 1-28 of treatment period.
  Interventions: Drug: Placebo
- 2 (Ramelteon) (Active Comparator): Patients will take 8 mgs of ramelteon 30 minutes before bedtime days 1-28 of treatment period.
  Interventions: Drug: Ramelteon

INTERVENTIONS:
Drug: Placebo — Placebo taken 30 minutes before bedtime days 1-28 of treatment period
  Arms: 1 (Placebo)
Drug: Ramelteon — 8 mgs daily for days 1-28 of treatment period
  Other Names: Rozerem
  Arms: 2 (Ramelteon)

SUMMARY:
This study is being conducted to evaluate the effectiveness of ramelteon 8mgs in the treatment of insomnia in patients that have completed their first chemotherapy treatment for breast cancer.

DETAILED DESCRIPTION:
Phase IV, randomized, double-blind, placebo-controlled, parallel-group study to assess the efficacy of ramelteon 8mgs in the treatment of insomnia in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 21-60 years old
* Have a negative serum or urine pregnancy test for women of child-bearing potential
* Have a three-month or longer history of insomnia
* Self-report < 6.5 hours of total sleep time, in addition to a sleep efficiency of less than 85%, averaged over two weeks of screening
* A score of less than 60 on the Zung Self-Rating Depression Scale
* Self-report bedtimes that do not vary by more than two hours on five nights per week
* Have completed chemotherapy for breast cancer less than two years prior to study drug administration
* Have completed chemotherapy for breast cancer for at least two months prior to screening visit
* Patients that are receiving Herceptin are eligible for study enrollment
* Have completed radiation therapy for breast cancer for at least two months prior to screening visit
* ECOG (Eastern Cooperative Oncology Group)score of 0-1
* Be able to read, understand, and provide written informed consent before enrolling in the study
* Must be willing to comply with all study visits and comply with daily phone calls to the IVRS throughout the study
* Agree to participate for the entire study period (about two months)

Exclusion Criteria:

* Metastatic disease
* Pregnant or lactating female
* Self-reports typical consumption of more than five alcoholic beverages on a single day or greater than 14 alcoholic beverages weekly
* Self-reports use of products containing nicotine of greater than 15 cigarettes daily or cannot avoid products containing nicotine during sleep periods
* Current use of any of the following medications, and cannot discontinue these medications for the duration of the study: Hypnotic medication, Anti-convulsants, Anxiolytics, Narcotic analgesics, Medications or supplements containing Melatonin, Ketaconazole and Fluconazole
* Currently taking fluvoxamine, brand name Luvox
* Have symptoms consistent with the diagnosis of any other sleep disorder other than insomnia (e.g. obstructive sleep apnea, narcolepsy, restless legs syndrome)
* Currently on night or rotating shift work
* Self-reports habitual napping of greater than one hour accumulated sleep on 4 or more days per week
* Has a psychiatric illness that interferes with normal sleep-wake function (e.g. major depression, post-traumatic stress disorder)
* A score of 60 or greater on the Zung Self-Rating Depression Scale
* Has current unstable medical disorder, such as symptomatic congestive heart failure, uncontrolled cardiac arrhythmia, or other serious medical condition as determined by the Investigator

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-08; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward J. Stepanski, Ph.D., Study Chair — Accelerated Community Oncology Research Network
Locations (10):
- United States (10):
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Wilshire Oncology Medical Group, Inc., La Verne, California
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Augusta Oncology Associates, PC, Augusta, Georgia
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Hematology Oncology Centers of the Northern Rockies, Billings, Montana
  - Tri-County Hematology & Oncology Associates, Canton, Ohio
  - Pottsville Cancer Center, Pottsville, Pennsylvania
  - The West Clinic, Memphis, Tennessee
  - Cancer Specialists of Tidewater, Ltd., Chesapeake, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 community oncology research sites across the United States within Accelerated Community Oncology Research Network (ACORN) participated in this study. Enrollment started in August 2006 and closed in August 2008.
Pre-assignment Details: After consent, subjects underwent a 2 week screening period to see if they met the criteria for insomnia and to assess compliance with daily Interactive Voice Recognition System (IVRS) calls.
Period: Screening Period (Pre-randomization)
Arm/Group | 1 (Placebo) | 2 (Ramelteon)
Started | 22 (22 subjects were consented. All subjects received placebo during the 2 week screening period.) | 0
Completed | 16 (16 subjects completed the screening period and were eligible for randomization.) | 0
Not Completed | 6 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Non-compliance | 1 | 0
Not completed — Screen failure | 3 | 0
Period: Treatment Period
Arm/Group | 1 (Placebo) | 2 (Ramelteon)
Started | 7 (16 subjects were randomized to either placebo or ramelteon before starting treatment period.) | 9 (16 subjects were randomized to either placebo or ramelteon before starting treatment period.)
Randomization | 7 | 9
Completed | 6 | 7
Not Completed | 1 | 2
Not completed — Non-compliance | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Withdrawal Period
Arm/Group | 1 (Placebo) | 2 (Ramelteon)
Started | 6 (Subjects in both groups received placebo for one week.) | 7 (Subjects in both groups received placebo for one week.)
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 (Placebo) | 2 (Ramelteon) | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 51.69 (5.98) | 49.11 (6.78) | 50.24 (6.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency
Description: Total time in bed is calculated as the time the subject got out of bed minus the time the subject went to bed. The total sleep time is reported by the subject. Percent sleep efficiency is calulated as 100*(total sleep time divided by total time in bed).
Time Frame: Every morning during the screening, treatment, and withdrawal periods
Population: Screening period: 14 patients with 6 treated with Placebo and 8 with Ramelteon. Treatment period: 13 patients with 5 treated with Placebo and 8 with Ramelteon. Withdrawal period: 10 patients with 4 treated with Placebo and 6 with Ramelteon.
Measure: Mean (Standard Deviation); unit: Percent sleep efficiency
Arm/Group | 1 (Placebo) | 2 (Ramelteon)
Number analyzed (Participants) | 6 | 8
Percent sleep efficiency
  Screening Period | 59.62 (16.72) | 70.16 (12.55)
  Treatment Period | 72.09 (9.38) | 71.26 (14.54)
  Withdrawal Period | 75.87 (11.85) | 67.48 (14.19)

2. Secondary Outcome: Quantitative Sleep Parameters - Total Sleep Time
Description: The subject reports how many hours of sleep she got.
Time Frame: Every morning during the screening, treatment, and withdrawal periods
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 1 (Placebo) | 2 (Ramelteon)
Number analyzed (Participants) | 6 | 8
Hours
  Screening Period | 5.02 (1.62) | 5.27 (0.83)
  Treatment Period | 5.94 (1.20) | 5.62 (0.79)
  Withdrawal Period | 5.57 (0.50) | 5.11 (0.87)

3. Secondary Outcome: Quantitative Sleep Parameters - Number of Awakenings
Description: The subject reports how many times she woke up during the night.
Time Frame: Every morning during the screening, treatment, and withdrawal periods
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Awakenings
Arm/Group | 1 (Placebo) | 2 (Ramelteon)
Number analyzed (Participants) | 6 | 8
Awakenings
  Screening Period | 2.62 (0.46) | 2.66 (1.10)
  Treatment Period | 2.28 (0.37) | 2.76 (1.70)
  Withdrawal Period | 2.19 (1.18) | 2.37 (0.80)

4. Secondary Outcome: Qualitative Evaluation of Sleep - Global Sleep Impression
Description: The Patient Global Impression is a 7-point scale which asks "How much has your sleep improved?" with the following anchors: no improvement, minimal improvement, slight improvement, moderate improvement, very good improvement, near complete improvement, and complete improvement.
Time Frame: Once during the withdrawal period
Measure: Number; unit: Participants
Arm/Group | 1 (Placebo) | 2 (Ramelteon)
Number analyzed (Participants) | 6 | 7
Participants
  Complete improvement | 0 | 1
  Moderate improvement | 3 | 0
  Slight improvement | 1 | 0
  Minimal improvement | 0 | 2
  No improvement | 2 | 4

5. Secondary Outcome: Qualitative Evaluation of Sleep - Quality of Sleep
Description: The subject rates the quality of her sleep on a scale of 0 through 10, where 0 is a very bad night of sleep and 10 is a very good night of sleep.
Time Frame: Every morning during the screening, treatment, and withdrawal periods
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | 1 (Placebo) | 2 (Ramelteon)
Number analyzed (Participants) | 6 | 8
Units on a Scale
  Screening Period | 4.60 (1.32) | 5.32 (0.78)
  Treatment Period | 5.47 (1.25) | 5.15 (0.93)
  Withdrawal Period | 6.59 (2.06) | 5.47 (0.68)

6. Secondary Outcome: Daytime Function - Fatigue
Description: The subject rates her fatigue on a scale of 0 through 10, where 0 is not a problem and 10 is as bad as possible.
Time Frame: Once during the screening period; once during the treatment period; twice during the withdrawal period for a total of 4 assessments
Population: Screening period: 12 patients with 6 treated with Placebo and 6 with Ramelteon. Treatment period: 11 patients with 4 treated with Placebo and 7 with Ramelteon. Withdrawal period: 8 patients with 4 treated with Placebo and 4 with Ramelteon.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | 1 (Placebo) | 2 (Ramelteon)
Number analyzed (Participants) | 6 | 6
Units on a Scale
  Screening Period | 3.06 (2.36) | 2.11 (1.70)
  Treatment Period | 2.42 (0.79) | 4.07 (1.84)
  Withdrawal Period | 3.38 (2.43) | 3.00 (2.45)

7. Secondary Outcome: Daytime Function - Despair
Description: The subject rates 7 questions related to despair on a scale of 0 through 10 for each question, where 0 is not bad and 10 is as bad as possible. The scores of these 7 questions are combined and normalized, and used to describe despair.
Time Frame: as for outcome 6
Population: Screening period: 11 patients with 6 treated with Placebo and 5 with Ramelteon. Treatment period: 9 patients with 4 treated with Placebo and 5 with Ramelteon. Withdrawal period: 8 patients with 4 treated with Placebo and 4 with Ramelteon.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | 1 (Placebo) | 2 (Ramelteon)
Number analyzed (Participants) | 6 | 5
Units on a Scale
  Screening Period | 47.07 (10.17) | 46.02 (6.92)
  Treatment Period | 42.92 (0.00) | 45.15 (5.00)
  Withdrawal Period | 49.38 (12.91) | 42.92 (0.00)

8. Secondary Outcome: Daytime Function - Distress
Description: The subject rates 4 questions related to distress on a scale of 0 through 10 for each question, where 0 is not bad and 10 is as bad as possible. The scores of these 4 questions are combined and normalized, and used to describe distress.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | 1 (Placebo) | 2 (Ramelteon)
Number analyzed (Participants) | 6 | 5
Units on a Scale
  Screening Period | 42.91 (12.20) | 41.99 (9.07)
  Treatment Period | 37.93 (0.00) | 39.86 (4.32)
  Withdrawal Period | 45.40 (14.94) | 37.93 (0.00)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected beginning at Visit 2: Randomization Visit (Day 1) until Visit 4: Close-out Visit (Day 36).
Description: Systematic Assessment - subjects were assessed for adverse events at each study visit by either the research coordinator, treating physician, or other appropriate sub-investigator (such as a nurse practitioner or physician assistant).
Arm/Group | 1 (Placebo) | 2 (Ramelteon)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 6/7 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 (Placebo) (N=7) | 2 (Ramelteon) (N=9)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Leg edema (General disorders) | 1 (1) | 0 (0)
Pain on right side of chest (General disorders) | 1 (1) | 0 (0)
Abscess on right hip (Infections and infestations) | 1 (1) | 1 (1)
Sinus infection (Infections and infestations) | 0 (0) | 1 (1)
Yeast infection (Infections and infestations) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Coughing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory virus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early study termination due to slow enrollment; Small sample size analyzed; Some IVRS and Patient Care Monitor (PCM) data were lost and could not be retrieved; Some subject non-compliance with study requirements

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must provide Sponsor an advance copy of any proposed publication whether in journals or in conferences or other public forum at least 60 days prior to any submission for publication or public presentation so that Sponsor may determine whether it contains any Confidential Information of Sponsor, and/or any discovery or invention is made.